CLINICAL TRIAL: NCT00074867
Title: A Clinical Efficacy Study Of An Oral Tyrosine Kinase Inhibitor Of VEGFR-2 To Treat Recurrent Or Persistent Small-Volume Epithelial Ovarian Cancer, Primary Peritoneal Serous Cancer, Or Fallopian Tube Cancer
Brief Title: Study Of An Oral Tyrosine Kinase Inhibitor Of VEGFR-2 To Treat Small-Volume Ovarian, Peritoneal, Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3521003
Record Dates: First submitted 2003-12-22; First posted 2003-12-24 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-07

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms | interventions — 3-(4-bromo-2,6-difluorobenzyloxy)-5-(3-(4-pyrrolidin-1-ylbutyl)ureido)isothiazole-4-carboxylic acid amide

INTERVENTIONS:
Drug: CP-547,632

SUMMARY:
The purpose of this study is to determine whether CP-547,632, an oral VEGFR-2 tyrosine kinase inhibitor is effective in the treatment of epithelial ovarian cancer, primary peritoneal serous cancer, or fallopian tube cancer for patients who have failed first line platinum-based therapy and have a persistent rising CA-125.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven epithelial ovarian cancer, primary peritoneal serous cancer, or fallopian tube cancerRecurrent or persistent elevated CA-125.
* For the purpose of this study, elevated CA-125 is defined as a value of â‰¥40 U/ml on two separate consecutive determinations made â‰¥1 week apart.
* CA-125 values obtained within 4 weeks of abdominal surgery should not be taken into account.
* No definitive disease or clinical and findings of small volume disease (£1cm by spiral CT or £2cm by conventional CT or clinical exam).

Exclusion Criteria:

* No prior exposure to mouse antibodies or prior VEGF or VEGF receptor targeted treatment or other anti-angiogenic-directed, anti-cancer treatment including thalidomide.
* No prior consolidation therapy with cytotoxic agents for ovarian cancer.
* Continuation of hormone replacement therapy is permitted.
* No requirement for concomitant anticoagulant therapy.
* Administration of low dose anticoagulants for maintenance of central venous access is permitted.No chronic oral or intravenous steroid use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29
Dates: Start 2003-10; Study Completion 2004-09

PRIMARY OUTCOMES:
At the completion of Stage 1 of the study, it did not meet the objective response criteria to proceed to Stage 2 of the trial.

SECONDARY OUTCOMES:
Given the outcome of the primary objective, analysis of secondary objectives were not formalized.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (5):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, New York, New York
- Canada (2):
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Québec, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3521003&StudyName=Study+Of+An+Oral+Tyrosine+Kinase+Inhibitor+Of+VEGFR%2D2+To+Treat+Small%2DVolume+Ovarian%2C+Peritoneal%2C+Fallopian+Tube+Cancer+